CLINICAL TRIAL: NCT00061100
Title: HIV Counseling Intervention for Methadone-Maintained Patients
Brief Title: HIV Counseling Intervention for Methadone-Maintained Patients - 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #3884; R01DA011444 (NIH); 3884 (Other: NYSPI IRB)
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Opioid-Related Disorders
Keywords: HIV; methadone maintenance
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RISE intervention (Experimental): Targeted RISE intervention- Behavior therapy Rise
  Interventions: Behavioral: Behavior Therapy-RISE
- Standard Education (Active Comparator): Education intervention. Standard prevention education
  Interventions: Behavioral: Standard prevention Education

INTERVENTIONS:
Behavioral: Behavior Therapy-RISE — manually-guided HIV intervention RISE: Reduce high risk Intravenous drug use and unsafe Sexual Encounter
  Arms: RISE intervention
Behavioral: Standard prevention Education — standard psychosocial Education for HIV/hepatitis prevention
  Arms: Standard Education

SUMMARY:
The purpose of this study is to evaluate HIV counseling intervention for Methadone-Maintained Patients.

DETAILED DESCRIPTION:
The purpose of this proposal is to evaluate, in methadone-maintained patients the association between an ADHD diagnosis and high-risk HIV/Hepatitis behavior. In addition, the investigators would like to determine whether a new manually-guided HIV intervention; RISE: Reduce high risk Intravenous drug use and unsafe Sexual Encounters is superior to standard HIV/Hepatitis psycho-education.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM-IV criteria for opiate dependence and currently in methadone maintenance treatment
* Able to give informed consent and capable of complying with study procedures
* Women who are of childbearing age and/or pregnant may be included
* Individuals who are HIV-positive or have Acquired Immunodeficiency Syndrome may be included
* Patients who demonstrate moderate to high HIV risk behaviors will be included
* Patients with low to no HIV risk behaviors will be excluded
* Patients receiving a stable dose of methadone for three weeks will be included

Exclusion Criteria:

* Currently meets DSM-IV criteria for current Axis I psychiatric disorders (other than ADHD or substance abuse) which requires medical intervention, i.e., active suicide ideation, active psychosis, anxiety disorders, depression requiring hospitalization
* Patients who have exhibited suicidal or homicidal behavior within the past two years
* HIV positive patients must have knowledge of their status for a minimum of three weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 1999-10; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
AIDS risk behavior based on the Risk Behavior Assessment | assessed monthly during 2 months of study or length of participation

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- Research Foundation for Mental Hygiene, Inc., New York, New York, United States